CLINICAL TRIAL: NCT05571319
Title: Study of Metformin to Reduce Cerebrovascular Dysfunction in South African Patients With HIV and Metabolic syndRome: a Pilot Trial.
Brief Title: A Pilot Study of Metformin to Reduce Cerebrovascular Dysfunction in Participants With HIV and Metabolic Syndrome.
Acronym: SMART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Collaborators: University of Rochester (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Eric Decloedt, Associate Professor & Head of Clinical Pharmacology, University of Stellenbosch
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21/10/024; R21TW012185-01 (NIH)
Record Dates: First submitted 2022-06-28; First posted 2022-10-07 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Syndrome; HIV Seropositivity
Keywords: pilot open label trial; cerebrovascular dysfunction; endothelial function
MeSH Terms: conditions — Metabolic Syndrome; HIV Seropositivity

STUDY DESIGN:
Intervention Model Description: We will enroll 30 participants in an open-label study of metformin treatment for 12 weeks with a 4-week washout period and a final evaluation. The 4-week washout period was chosen to assess the post-treatment effect of metformin on peripheral markers of endothelial function, with expectation that those measurements will trend toward the baseline values.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label arm (Experimental): All participants to receive metformin extended-release 1000mg to 2000mg daily for 12 weeks.
  Interventions: Drug: Metformin Extended Release Oral Tablet

INTERVENTIONS:
Drug: Metformin Extended Release Oral Tablet — Glucophage XR 500 mg

SUMMARY:
Metabolic syndrome is a constellation of risk factors for cardiovascular disease and type 2 diabetes mellitus which frequently occur together. Data is emerging suggesting metabolic syndrome causes brain disease by contributing to blood vessel damage and inflammation. People living with HIV (PLWH) are at high risk and the investigators will perform a pilot study of the well-known type 2 diabetes drug metformin to treat this blood vessel damage and inflammation in PLWH.

DETAILED DESCRIPTION:
Background: Metabolic syndrome (MetS) is a constellation of risk factors for cardiovascular disease and type 2 diabetes mellitus (T2D) which frequently occur together. The consequences of MetS extend beyond the increased risk of vascular-metabolic disease. Data is emerging suggesting causality between MetS and cerebral small vessel disease. MetS is associated with an increased incidence of vascular dementia and progression from mild cognitive impairment to dementia. MetS cause endothelial dysfunction and low-level inflammation of adipose tissue. MetS-associated endothelial dysfunction is independent of obesity status with an increased number of MetS abnormalities correlating with more endothelial dysfunction. Middle cerebral artery stiffening with impaired blood flow is associated with a higher MetS score.

Enhanced access to effective combination antiretroviral therapy (cART) improved the life expectancy of people living with HIV (PLWH) substantially. Longevity, however, presents unique health challenges, one being the development of non-communicable diseases including MetS. Emerging data from sub-Saharan Africa indicate a higher prevalence of MetS among PLWH compared with their HIV-negative counterparts. The incidence of MetS in PLWH is predicted to increase. Abdominal obesity is reaching alarming proportions in sub-Saharan Africa with the prevalence similar to that of high-income countries. Older antiretroviral regimens are associated with higher treatment-emergent MetS. Given the growing HIV-positive population with MetS, and that both MetS and HIV are chronic inflammatory conditions, there is an urgent need to identify effective and affordable pharmacotherapy that addresses modifiable aspects of vascular disease.

The investigtors hypothesise that metformin is effective in treating endothelial dysfunction and thus ameliorating cerebrovascular function in HIV-positive patients with metabolic syndrome. Metformin has been shown to affect endothelial cells by inhibiting several inflammatory molecules. Pilot clinical trial data support that metformin significantly improves endothelial function, even in short-term treatment. Metformin is a low-cost and well-known drug used for the management of abnormal glucose homeostasis in people with T2D. Metformin is widely available in public service settings and is considered to have a clinical effect beyond glucose lowering. Based on the rationale above, the investigators propose to study metformin in HIV-positive participants with MetS who are virologically suppressed by standard of care cART to receive open-label metformin to assess its effect on cerebrovascular function.

Objective: The investigators propose to address the Specific Aims listed below in HIV-positive participants with metabolic syndrome virologically suppressed on standard of care cART receiving open-label metformin 12 weeks. Aim 1: To obtain preliminary data on the effect of metformin on cerebral vascular reactivity and cerebral blood flow in HIV positive participants with metabolic syndrome. Aim 2: To assess whether metformin associated changes in cerebral vascular reactivity and cerebral blood flow (CBF) are mediated via improvements in endothelial function.

Methods: The investigators will enroll 30 participants in an open-label study of metformin treatment for 12 weeks with a 4-week washout period and a final evaluation. Comprehensive metabolic, laboratory and neuroimaging evaluation will be performed at screening and 12 weeks with selected procedures repeat after the 4 weeks washout period at week 16. Whole body dual-energy X-ray absorptiometry (DEXA) at study entry will be used to assess adipose tissue location.

Outcome: The purpose of this pilot study in PLWH with MetS is to obtain preliminary data on the effect of metformin on cerebrovascular function using non-invasive neuroimaging biomarkers. Furthermore, the investigators will test the hypothesis that metformin mediates the cerebrovascular changes in part via endothelial regulation by using a comprehensive panel of endothelial functional and soluble markers which will be correlated with the imaging metrics. The results of the study will form the basis for a future clinical trial that will assess the beneficial effect of metformin in reducing the burden of cerebral small vessel disease in PLWH.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years);
* HIV+ on antiretroviral therapy for at least 12 months prior to study entry;
* Viral load ≤50 copies/mL;
* Able to provide informed consent;
* Metabolic syndrome as per the harmonized criteria;
* Women of child-bearing potential willing to use adequate contraception (defined as either an intra-uterine contraceptive device or hormonal contraceptive);

Exclusion Criteria:

* Treated with metformin as part of care;
* History of drug or alcohol abuse within 3 months before screening;
* Known neurosyphilis;
* Known vitamin B12 deficiency;
* Known neuropsychiatric disorders or serious psychiatric symptoms;
* Significant head trauma with imaging structural abnormalities;
* Renal impairment (estimated glomerular filtration < 60 mL/min/1.73m2);
* Type I or type II diabetes (fasting plasma glucose >7mmol/L and/or HbA1c >6.5%);
* Hypersensitivity to metformin;
* Any contraindication or special precaution in the metformin package insert which may put the participant at a safety risk;
* Cationic drugs (as listed in the metformin package insert) that may increase metformin concentrations significantly;
* Claustrophobia, metal implants or any other condition that prevents performing MR scan;
* Pregnant / breastfeeding;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Outcome: cerebral reactivity. | 12 weeks
  We will measure changes in cerebrovascular reactivity (percentage change of BOLD signal during resting state fMRI) from baseline to 12 weeks.
Outcome: cerebral blood flow. | 12 weeks
  We will measure changes in cerebral blood flow (mL/100mL/min, via arterial spin labeling) from baseline to 12 weeks.
Outcome: peripheral vascular reactivity. | 12 weeks
  We will measure changes in finger reactive hyperemia index from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Decloedt, MBChB, PhD, Principal Investigator — University of Stellenbosch
Locations (1):
- Desmond Tutu Health Foundation: Gugulethu Research Site, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The raw study data will be made available to individuals or organisations who make legitimate and appropriate requests, provided that permission from the collaborators and their institutions, sponsor, funder and the Stellenbosch University Human Research Ethics Committee have been obtained.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within10 working days after all the permissions have been obtained.
Access Criteria: Legitimate and appropriate requests (as evaluated by the investigators, sponsor, funder and ethics committee).